CLINICAL TRIAL: NCT00759967
Title: Randomized Cross-over Study of Short Daily Hemodialysis Compared to Conventional Hemodialysis to Determine the Mechanisms of Hypertension Control
Brief Title: Conventional Hemodialysis vs. Short Daily Hemodialysis (6 Days / Week) and Mechanisms of Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other); University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2006 77401H
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-01

CONDITIONS: End Stage Renal Disease
Keywords: Randomized; Cross-Over; Conventional; Daily; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Catecholamines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short daily hemodialysis (Active Comparator): After a 3 month run-in period patients who are randomized to this arm will receive 3 months of short daily hemodialysis(2 hours/day,6 days/week)B/P will be monitored according to the Canadian hypertension guidelines both pre and post each dialysis session. Antihypertensive medication will be adjusted accordingly to maintain BP within the guidelines.At the end of this 3 month period extracellular fluid volume (bioimpedance) will be measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress will be collected.
  Interventions: Procedure: Microneurography; Procedure: Bioimpedance testing
- Conventional hemodialysis (Active Comparator): After a 3 month run-in period patients who are randomized to this arm will receive 3 months of conventional hemodialysis 3 days/week 3.5-4 hours/ treatment. BP will be monitored according to the Canadian hypertension guidelines both pre and post each dialysis session. Antihypertensive medication will be adjusted accordingly to maintain BP within the guidelines.At the end of this 3 moth period extracellular fluid volume (bioimpedance) will be measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress will be collected.
  Interventions: Procedure: Microneurography; Procedure: Bioimpedance testing

INTERVENTIONS:
Procedure: Microneurography — Muscle sympathetic nerve activity measurement will be obtained using microneurography. Approximately 10-20% of microneurography recordings are not interpretable due to technical problems. For this reason, blood samples will be collected at the same time that the microneurography is to be done. These test will be done at 3 time points throughout the study.
  Other Names: Catecholamines
Procedure: Bioimpedance testing — bioimpedance measurement of extracellular fluid volume will be measured at the end of each 3 month period. This test will be done at 3 time points throughout the study.
  Other Names: Bioimpedance; extracellular fluid volume measurement

SUMMARY:
More than 80% of patients with end stage renal disease have hypertension; 70% of whom are poorly controlled using conventional Hemodialysis therapy. An expanded extracellular fluid volume and an increase in peripheral vascular resistance as a result of hemodynamic/trophic effects of an increased sympathetic nerve activity, angiotensin II, asymmetrical dimethyl arginine, and decreased nitric oxide are the most frequently quoted mechanisms contributing to hypertension in this population. The intermittent nature of conventional hemodialysis treatments (4 hours, 3 days/week) results in the majority of patients having a sustained expansion of the extracellular fluid volume that likely contributes to the activation of neurohormonal pathways. However, daily therapy including short daily hemodialysis (2 hours, 6 days/week) and nocturnal hemodialysis (6-8 hours, 5-6 days/week) improve or even normalize blood pressure. Short daily hemodialysis appears to improve blood pressure secondary to a reduction in extracellular fluid volume (7,8) whereas the improvement in blood pressure with nocturnal hemodialysis occurs by a reduction in peripheral vascular resistance (8,9,10). This is consistent with the Katzarski et al experience (7-8 hours, 3 days/week) and one randomized controlled trial in which blood pressure control was due to normalization of extracellular fluid volume in some patients and a reduction in peripheral vascular resistance in others. The majority of the studies in daily dialysis are observational, do not include a run-in period to optimize blood pressure management and have not explored the mechanisms of improvement in blood pressure in detail. We have designed a 9 month study to determine if the mechanism by which short daily hemodialysis is associated with an improvement in blood pressure control is secondary to changes in sympathetic nervous system activity and/ or extracellular fluid volume. Additionally we would like to explore the potential impact of short daily dialysis, compared to conventional dialysis, on markers of inflammation and oxidative stress in detail.

DETAILED DESCRIPTION:
Patients with end stage renal disease have an adjusted risk of cardiovascular mortality that is 10-20 times greater than the general population. Of the modifiable risk factors, hypertension occurs in 80% of patients with end stage renal disease and is poorly controlled in 70% of patients. In several observational studies of daily hemodialysis, blood pressure has improved despite a reduction in the number of antihypertensive medications. A randomized crossover study in short daily hemodialysis also showed an improvement in systolic blood pressure and a reduction in left ventricular mass index. In limited investigation, the mechanism(s) responsible for the improvement in blood pressure have been attributed to a reduction in extracellular fluid volume (short daily) and a reduction in peripheral vascular resistance (nocturnal hemodialysis). The studies to date have been limited by failing to include a run in phase to optimize extracellular fluid volume prior to the initiation of daily dialysis. Additionally, only one study used a standardized algorithm for the management of blood pressure which is vital as the treatments are not blinded. We have designed a randomized, unblinded, 9 month cross-over study to determine the mechanism of blood pressure control on patients receiving conventional (3 times /week) HD to short daily HD (6 times /week 2 hrs/tx). After completing a 3 month run-in phase on conventional HD in which patient's dry weight and antihypertensive medications will be adjusted using a standardized algorithm, patients are to be randomized to a 3 month cross-over of daily HD versus conventional HD. The mechanism of improved blood pressure control will be explored using bioelectrical impedance to measure extracellular fluid volume (ECFV) and muscle sympathetic nerve activity (MSNA) as well as plasma catecholamines to measure the activity of the sympathetic nervous system. Additionally the effect of short daily HD, compared to conventional HD, on reactive oxygen species and markers of inflammation will be examined in Dr. Rhian Touyz lab. Lastly we will determine the patient's treatment preference.

ELIGIBILITY:
Inclusion Criteria:

* Systolic Hypertension
* They are able to make the time commitment for daily therapy
* They are capable of giving informed consent.

Exclusion Criteria:

* They are expected to receive a transplant within the next 12 months
* If they are considering a switch to peritoneal dialysis
* They are not expected to survive 12 months
* They have infections that require isolation (Vancomycin Resistant Enterococcus, Methicillin Resistant Staphylococcus Aureus, Hepatitis B)
* They have known symptomatic dilated cardiomyopathy (New York Association Class II or III with left ventricle ejection fraction of <0.35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Zimmerman, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Zimmerman DL, Ruzicka M, Hebert P, Fergusson D, Touyz RM, Burns KD. Short daily versus conventional hemodialysis for hypertensive patients: a randomized cross-over study. PLoS One. 2014 May 29;9(5):e97135. doi: 10.1371/journal.pone.0097135. eCollection 2014. PMID 24875804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 patients were recruited from the hemodialysis (HD) units of the Ottawa Hospital. 3 patients withdrew prior to randomization. 19 patients complete the conventional arm of the study, 2 patients withdrew during the short daily HD arm - they are included in the intention to treat analysis
Pre-assignment Details: There was a 3 month run in phase in which blood pressure was optimized prior to randomization. The 3 patients who were not randomized - 1) withdrew consent, he did not want his blood pressure taken routinely in dialysis, 2) one patient had concerns about medications being removed during daily dialysis that could not be reconciled, 3) screen failure
Groups:
- Conventional Hemodialysis First, Then Short Daily Hemodialysis: After a 3 month run-in period patients who are randomized to this arm received 3 months of conventional hemodialysis 3 days/week 3.5-4 hours/ treatment. BP was monitored according to the Canadian hypertension guidelines both pre and post each dialysis session. Antihypertensive medication were adjusted accordingly to maintain BP within the guidelines. At the end of this 3 moth period, extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress were collected.
  In this group 10 participants started and completed the first intervention: Conventional Hemodialysis first (Period Table 1; Left Column). These 10 participants then started the second intervention: Short Daily Hemodialysis (Period Table 2: Left Column), of which 8 participants completed the Short Daily Hemodialysis.
- Short Daily Hemodialysis First, Then Conventional Hemodialysis: After a 3 month run-in period patients who were randomized to this arm received 3 months of short daily hemodialysis(2 hours/day,6 days/week). Blood pressure was monitored according to the Canadian hypertension guidelines both pre and post each dialysis session. Antihypertensive medication was adjusted accordingly to maintain BP within the guidelines. At the end of this 3 month period, extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress were collected.
  In this group 9 participants started and completed the first intervention: Short Daily Hemodialysis first (Period Table 1: Right Column). These 9 participants then started the second intervention: Conventional Hemodialysis (Period Table 2: Right Column). All 9 participants finished conventional dialysis.
Period: First Intervention
Arm/Group | Conventional Hemodialysis First, Then Short Daily Hemodialysis | Short Daily Hemodialysis First, Then Conventional Hemodialysis
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Conventional Hemodialysis First, Then Short Daily Hemodialysis | Short Daily Hemodialysis First, Then Conventional Hemodialysis
Started | 10 | 9
Completed | 8 | 9
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: 3 patients withdrew prior to randomization, analysis based on the 19 patients randomized
Groups:
- All Participants: All patients in the study were randomized after the 3 month run in phase to either Conventional HD or Short Daily HD for 3 months and then crossed over to the other treatment arm for 3 months
Arm/Group | All Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Region of Enrollment [Number; unit: participants]
  Canada | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Systolic Blood Pressure Over the Third Month of Each Treatment Arm
Description: The average of 2 measurements taken pre each dialysis session in the third month of treatment were compared when the patients were on conventional hemodialysis compared to short daily hemodialysis. SBP was taken in accordance with guidelines from the Canadian Hypertension Society
Time Frame: Average of the last month of the 3 month intervention
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Short Daily Hemodialysis: After a 3 month run-in period patients who were randomized to this arm received 3 months of short daily hemodialysis(2 hours/day,6 days/week). SBP was monitored according to the Canadian hypertension guidelines pre each dialysis session. Antihypertensive medication was adjusted accordingly to maintain BP within the guidelines. At the end of the 3 moth period extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress were collected.
- Conventional Hemodialysis: After a 3 month run-in period patients randomized to this arm received 3 months of conventional hemodialysis 3 days/week 3.5-4 hours/ treatment. SBP was monitored according to the Canadian hypertension guidelines pre each dialysis session. Antihypertensive medication was adjusted accordingly to maintain BP within the guidelines. At the end of this 3 moth period extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress were collected.
Arm/Group | Short Daily Hemodialysis | Conventional Hemodialysis
Number analyzed (Participants) | 19 | 19
mm Hg | 139 (14) | 142 (17)

2. Secondary Outcome: To Determine if the Mechanism by Which Short Daily Hemodialysis is Associated With Changes in Extracellular Fluid Volume
Description: The extracellular fluid volume will be measured using bioelectrical impedance to determine if the mechanism by which short daily hemodialysis is associated with an improvement in blood pressure control is secondary to changes in extracellular fluid volume.
Time Frame: once the final participant has completed all intervention procedures, approx. 3 months
Measure: Mean (Standard Deviation); unit: Litres
Groups:
- Short Daily Hemodialysis: After a 3 month run-in period patients who were randomized to this arm received 3 months of short daily hemodialysis(2 hours/day,6 days/week). SBP was monitored according to the Canadian hypertension guidelines pre each dialysis session. Antihypertensive medication was adjusted accordingly to maintain BP within the guidelines. At the end of the 3 moth period extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress were collected.
  Below shows the results of the extracellular fluid volume
- Conventional Hemodialysis: After a 3 month run-in period patients randomized to this arm received 3 months of conventional hemodialysis 3 days/week 3.5-4 hours/ treatment. SBP was monitored according to the Canadian hypertension guidelines pre each dialysis session. Antihypertensive medication was adjusted accordingly to maintain BP within the guidelines. At the end of this 3 moth period extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress were collected.
  Below shows the results of the extracellular fluid volume
Arm/Group | Short Daily Hemodialysis | Conventional Hemodialysis
Number analyzed (Participants) | 19 | 19
Litres | 15.4 (2.8) | 15.2 (3.2)

3. Secondary Outcome: To Determine if Short Daily Hemodialysis, Compared to Conventional Hemodialysis Maintains Metabolic Homeostasis
Description: Serum phosphate values from the end of the three month run in phase and after randomization used to measure metabolic homeostasis
Time Frame: once the last participant has completed run in phase and after randomization, approx. 3 months
Measure: Mean (Standard Deviation); unit: mmol/Litre
Arm/Group | Short Daily Hemodialysis | Conventional Hemodialysis
Number analyzed (Participants) | 19 | 19
mmol/Litre
  Serum Phosphate at end of 3 month run-in phase | 1.61 (0.53) | 1.61 (0.53)
  Serum phosphate after randomization | 1.58 (0.41) | 1.82 (0.65)

4. Secondary Outcome: To Determine if the Enhance Control of Blood Pressure With Daily Hemodialysis Compare to Conventional Hemodialysis is Associated With a Reduction in Oxidative Stress.
Time Frame: once the final participant has completed all intervention procedures, approx. 3 months
Measure: Median (Inter-Quartile Range); unit: mmol/ml MDA equivalent
Groups:
- Short Daily Hemodialysis First, Then Conventional Hemodialysis: After a 3 month run-in period patients who were randomized to this arm received 3 months of short daily hemodialysis(2 hours/day,6 days/week). SBP was monitored according to the Canadian hypertension guidelines pre each dialysis session. Antihypertensive medication was adjusted accordingly to maintain BP within the guidelines. At the end of the 3 month period extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress were collected.
- Conventional Hemodialysis First, Then Short Daily Hemodialysis: After a 3 month run-in period patients randomized to this arm received 3 months of conventional hemodialysis 3 days/week 3.5-4 hours/ treatment. SBP was monitored according to the Canadian hypertension guidelines pre each dialysis session. Antihypertensive medication was adjusted accordingly to maintain BP within the guidelines. At the end of this 3 month period extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress were collected.
Arm/Group | Short Daily Hemodialysis First, Then Conventional Hemodialysis | Conventional Hemodialysis First, Then Short Daily Hemodialysis
Number analyzed (Participants) | 12 | 12
mmol/ml MDA equivalent
  TBARS Baseline | 2.3 [1.9 to 2.9] | 2.3 [1.9 to 2.9]
  TBARS After Randomization | 2.0 [1.7 to 3.1] | 2.4 [1.8 to 3.5]

5. Secondary Outcome: To Determine Patient Modality Preference.
Description: each participant will complete a questionaire regarding modality preference
Time Frame: at study completion
Population: The trial did not include a questionnaire regarding modality preference as originally planned
Arm/Group | Short Daily Hemodialysis | Conventional Hemodialysis
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: To Determine if the Enhance Control of Blood Pressure With Daily Hemodialysis Compare to Conventional Hemodialysis is Associated With a Reduction in Markers of Inflammation
Time Frame: once the final participant has completed all intervention procedures, approx. 3 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Short Daily Hemodialysis First, Then Conventional Hemodialysis | Conventional Hemodialysis First, Then Short Daily Hemodialysis
Number analyzed (Participants) | 12 | 12
pg/mL
  IL-6 Baseline | 1.55 [1.04 to 3.26] | 1.55 [1.04 to 3.26]
  IL-6 After Randomization | 1.52 [0.95 to 3.3] | 1.45 [0.65 to 3.08]

ADVERSE EVENTS:
Groups:
- Short Daily Hemodialysis: After a 3 month run-in period patients who are randomized to this arm received 3 months of short daily hemodialysis(2 hours/day,6 days/week). SBP was monitored according to the Canadian hypertension guidelines pre each dialysis session. Antihypertensive medication wer adjusted accordingly to maintain BP within the guidelines.At the end of this 3 moth period extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress will be collected.
- Conventional Hemodialysis: After a 3 month run-in period patients who were randomized to this arm received 3 months of conventional hemodialysis 3 days/week 3.5-4 hours/ treatment. SBP was monitored according to the Canadian hypertension guidelines pre each dialysis session. Antihypertensive medication was adjusted accordingly to maintain BP within the guidelines.At the end of this 3 moth period extracellular volume was measured using bioimpedance as well as sympathetic nerve activity using microneurography. Additionally Catecholamines as well as markers of oxidative stress were collected.
Arm/Group | Short Daily Hemodialysis | Conventional Hemodialysis
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Daily Hemodialysis (N=19) | Conventional Hemodialysis (N=19)
Hospitalization for congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) — Patient admitted to hospital for volume overload

LIMITATIONS AND CAVEATS:
Although 2 patients stopped doing short daily HD they were included in the intention to treat analysis with their short daily HD BPs carried forward

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No